CLINICAL TRIAL: NCT01064206
Title: Study of Psychological and Addictive Profile of Patients With Buerger's Disease
Brief Title: ADDICTAO: Psychological and Addictive Profile of Patients With Buerger's Disease
Acronym: ADDICTAO
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2008_03/0814; 2008-A00378-47 (Other: ID-RCB number, ANSM); PHRC 2008/1915 (Other: DHOS)
Record Dates: First submitted 2010-02-05; First posted 2010-02-08 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Thromboangiitis Obliterans; Atheromatous Arteritis
Keywords: thrombangiitis obliterans; Buerger's disease; atheromatous arteritis; psychiatric disorders; personality disorders; addictive profile; addiction; tobacco; cannabis
MeSH Terms: conditions — Thromboangiitis Obliterans; Mental Disorders; Personality Disorders; Behavior, Addictive; Marijuana Abuse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Buerger's disease patients: 200 thromboangiitis obliterans patients (Buerger's disease or TAO)
- Control group: 200 atheromatous arteritis patients

SUMMARY:
Background: Buerger's disease (thromboangiitis obliterans or TAO) is a rare disease (1/ 10 000) characterized by the development of segmental thrombotic occlusions of the medium and small arteries of the extremities. Afflicted patients are mostly young, male, inveterate tobacco (or cannabis) smokers who present with distal extremity ischemia, ischemic ulcers, of the toes or fingers. Large arteries are typically spared, as are the coronary, cerebral, and visceral circulations. Patients with TAO often suffer from severe ischemic pain and tissue loss culminating in minor and major limb amputation. Clinical diagnostic criteria generally include history of tobacco abuse; age of onset less than 50 years; infrapopliteal, segmental arterial occlusions with sparing of the proximal vasculature; frequent distal upper extremity arterial involvement (Raynaud's syndrome or digital ulceration); superficial phlebitis; and exclusion of arteriosclerosis, diabetes, true arteritis, proximal embolic source, and hypercoagulable states.

While the cause of Buerger's disease remains unknown, the disease onset and clinical course are inextricably linked to tobacco (or cannabis) abuse. Tobacco abstinence generally results in disease quiescence and remains the mainstay of treatment. For some unknown reason, clinicians observed that TAO patients rarely discontinue smoking even though amputation is usually the inevitable consequence and the only method available of controlling pain and ulceration. Few studies were realized and Hofer-Mayer and coll. found remarkable personality features comparing to coronary patients: TAO patients significantly changed their place of work more often, had more absenteeism from work, smoked more before the illness and continued to smoke more frequently during their illness, were more often single or divorced and had more conflicts in their relationships. Those facts led us to explore their psychopathology and their addictive profile.

Purpose: Search the prevalence of personality disorders in Buerger's patients who present with tobacco or cannabis smoking.

Hypothesis: Patients with Buerger's disease show remarkable personality features (psychological and addictive profile) which are vulnerability factors to stop smoking (tobacco or cannabis) compared to patients with atheromatous arteritis.

DETAILED DESCRIPTION:
We include 200 Buerger's disease patients and 200 atheromatous arteritis patients, smoking tobacco or cannabis. First visit explores psychiatric disorders with MINI DSM IV (Lecrubier et al 1997), personality disorders with SCID II (Structured Clinical Interview for DSM IV); Addictive profile and Substance Use (or abuse) is evaluated with specific questionnaires (Rapid Addictive Profile, Fagerström and Cannabis questionnaire); Neuropsychological tests (Frontal Assessment Battery at bedside Dubois et al 2000; Stroop test , Stroop 1935); clinical assessment of the illness (Buerger and Atheromatous arteritis); and psychoactive substance and cotinine detection in urine. A second visit one year later will be realized with same assessments.

ELIGIBILITY:
Inclusion Criteria:

* Buerger's disease patients or atheromatous arteritis patients
* Smoking tobacco or cannabis

Exclusion Criteria:

* Diabetic patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We include 200 Buerger's disease patients and 200 atheromatous arteritis patients, smoking tobacco or cannabis
Sampling Method: Non-Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2008-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
SCID personality disorders | 2013

SECONDARY OUTCOMES:
psychiatric disorders by MINI DSM-IV results | 2013
RAP Fagerström and Cannabis questionnaire total scores | 2013
Results of neuropsychological assessment | 2013

CONTACTS AND LOCATIONS:
Overall Officials: Olivier COTTENCIN, Principal Investigator — University Hospital, Lille
Locations (16):
- France (16):
  - University Hospital, Bordeaux, Bordeaux
  - University Hospital, Brest, Brest
  - University Hospital, Caen, Caen
  - University Hospital, Lille, Lille
  - University Hospital, Marseille, Marseille
  - University Hospital, Montpellier, Montpellier
  - University Hospital, Nancy, Nancy
  - University Hospital, Nantes, Nantes
  - Georges Pompidou European Hospital, Paris, Paris
  - Tenon Hospital, Paris, Paris
  - University Hospital, Rouen, Rouen
  - University Hospital, Strasbourg, Strasbourg
  - University Hospital, Toulouse, Toulouse
  - University Hospital, Tours, Tours
  - General Hospital, Valenciennes, Valenciennes
  - Paul Brousse Hospital, Villejuif, Villejuif

IPD SHARING:
Plan to Share IPD: No